CLINICAL TRIAL: NCT06246994
Title: Predictors of Mortality Among Ventilator Associated Pneumonia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hussien kilany, principal investigator, Assiut University
Other Study IDs: Predictors of vap mortality
Record Dates: First submitted 2024-01-17; First posted 2024-02-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this context, this study aims to explore the risk factors for mortality from VAP in respiratory ICU.

DETAILED DESCRIPTION:
Pneumonia is the most common infection treated within ICUs and carries significant mortality risk . Ventilator-associated pneumonia (VAP) is a specific form of nosocomial pneumonia occurring in patients greater than 48 hours after intubation and the initiation of mechanical ventilation .

VAP is considered a leading cause of morbidity and mortality among intensive care unit infections. Despite various preventive measures, the incidence of VAP remains high .

In studies, VAP-related mortality is 14-70% . It is contemplated that there are independent risk factors, increasing VAP-related mortality .

However, the question of which factors are associated with early or late mortality in patients with VAP diagnosis, remains unanswered. Early identification and understanding of the etiology of VAP in the ICU is essential to prevent mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:This study will enroll:

1. adult participants over 18 years old who had undergone mechanical ventilation for longer than 48 hours.
2. Only the first episode of VAP for each patient will be included.

Exclusion Criteria:

1. Patients who are less than 18 years old.
2. Pneumonia diagnosed before mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult participants over 18 years old who had undergone mechanical ventilation for longer than 48 hours. Only the first episode of VAP for each patient will be included.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Mortality rate at 28 days. | 28 days
  Evaluation of number of dead patients from vap wihin 28 days of infection and
Percentage of risk factors of VAP mortality. | 28 days
  Search for risk factors for mortality of vap wihin 28 days of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Magdy, assisst -professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vincent JL, Sakr Y, Singer M, Martin-Loeches I, Machado FR, Marshall JC, Finfer S, Pelosi P, Brazzi L, Aditianingsih D, Timsit JF, Du B, Wittebole X, Maca J, Kannan S, Gorordo-Delsol LA, De Waele JJ, Mehta Y, Bonten MJM, Khanna AK, Kollef M, Human M, Angus DC; EPIC III Investigators. Prevalence and Outcomes of Infection Among Patients in Intensive Care Units in 2017. JAMA. 2020 Apr 21;323(15):1478-1487. doi: 10.1001/jama.2020.2717. PMID 32207816
- [Result] Zhou XY, Ben SQ, Chen HL, Ni SS. A comparison of APACHE II and CPIS scores for the prediction of 30-day mortality in patients with ventilator-associated pneumonia. Int J Infect Dis. 2015 Jan;30:144-7. doi: 10.1016/j.ijid.2014.11.005. Epub 2014 Nov 12. PMID 25461659
- [Result] Arayasukawat P, So-Ngern A, Reechaipichitkul W, Chumpangern W, Arunsurat I, Ratanawatkul P, Chuennok W. Microorganisms and clinical outcomes of early- and late-onset ventilator-associated pneumonia at Srinagarind Hospital, a tertiary center in Northeastern Thailand. BMC Pulm Med. 2021 Jan 30;21(1):47. doi: 10.1186/s12890-021-01415-8. PMID 33516213
- [Result] John AO, Paul H, Vijayakumar S, Anandan S, Sudarsan T, Abraham OC, Balaji V. Mortality from acinetobacter infections as compared to other infections among critically ill patients in South India: A prospective cohort study. Indian J Med Microbiol. 2020 Jan-Mar;38(1):24-31. doi: 10.4103/ijmm.IJMM_19_492. PMID 32719205
- [Result] Zimmerman JE, Kramer AA, McNair DS, Malila FM, Shaffer VL. Intensive care unit length of stay: Benchmarking based on Acute Physiology and Chronic Health Evaluation (APACHE) IV. Crit Care Med. 2006 Oct;34(10):2517-29. doi: 10.1097/01.CCM.0000240233.01711.D9. PMID 16932234